CLINICAL TRIAL: NCT04199091
Title: Craniosacral Therapy Versus Progressive Muscle Relaxation as Self-help Strategies for Patients With Chronic Non-specific Back Pain: a Randomized Controlled Trial
Brief Title: Craniosacral Therapy as a Self-help Strategy for Patients With Chronic Non-specific Back Pain
Acronym: CRANIO4ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Responsible Party: Principal Investigator, Heidemarie Haller, Principal Investigator, Universität Duisburg-Essen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19-8759-BO
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain, Mechanical; Complementary Therapies; Progressive Muscle Relaxation
Keywords: Craniosacral Therapy; Low Back Pain, Chronic; Randomized Controlled Trial; Self-help
MeSH Terms: conditions — Low Back Pain; Bronchiolitis Obliterans Syndrome | interventions — galactosylceramide sulfotransferase; Autogenic Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The investigator who will perform the group assignment will have no contact to the study participants. The outcome assessors will be blinded to group allocation. Patients will partly be blinded to the group intervention: The will be told that they will receive one of two self-help therapies - one that focus on the relaxation of fasciae and the other that focus on the relaxation of muscles. The statistician who will perform the analyses will kept blind to the group intervention by renaming groups with numbers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Craniosacral self-help techniques (CST) (Experimental): The experimental group consists of 24 teaching units (TUs) à 45 minutes over 12 weeks. The course starts with an introductory day (8 TUs), followed by 6 practice evenings every two weeks (2 TUs each) and a final afternoon (4 TUs). The patients will also receive a script with theoretical CST basics and descriptions of the techniques, which should facilitate the correct practice at home.
  Interventions: Procedure: Craniosacral Therapy (CST) self-help techniques
- Progressive muscle relaxation (PMR) (Active Comparator): The active control group consists of 24 teaching units (TUs) à 45 minutes over 12 weeks. Every week patients will meet for 2 TUs. The patients will also receive a script with theoretical basics and descriptions of the PMR techniques, hich should facilitate the correct practice at home.
  Interventions: Procedure: Progressive Muscle Relaxation (PMR)

INTERVENTIONS:
Procedure: Craniosacral Therapy (CST) self-help techniques — Manual self-help techniques based on Craniosacral Therapy (group setting).
  Arms: Craniosacral self-help techniques (CST)
Procedure: Progressive Muscle Relaxation (PMR) — Progressive muscle relaxation according to Jacobsen (group setting).
  Arms: Progressive muscle relaxation (PMR)

SUMMARY:
Craniosacral Therapy (CST) is a non-manipulative, very gentle manual treatment method. Although the mechanisms of action have not yet been investigated sufficiently, initial clinical trials support CST efficacy/effectiveness in chronic pain disorders such as back pain, neck pain, and fibromyalgia. In clinical practice, therapists also report pain alleviating effects of CST self-help techniques, offered to patients within a group concept. Yet, the effectiveness of teaching CST self-help techniques to medical laypersons has not yet been scientifically investigated.

Therefore, this study aims at collecting quantifiable data on the effectiveness and safety of a CST self-help group concept, developed for patients with chronic non-specific low back pain. The intervention group will receive 24 lessons of education and practice in CST self-help techniques over 12 weeks, while the control group will receive the same amount of self-help (education and practice) in progressive muscle relaxation. Six and 12 months after randomization, longer-term effects will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Chronic non-specific / functional lower back pain for at least 3 months
* Functional impairment: minimal 11 and maximal 41 points on the ODI
* Willingness to participate in the group program and practice at home

Exclusion Criteria:

* Specific back pain due to:
* Severe congenital or acute degenerative diseases
* Severe inflammatory musculoskeletal or rheumatic diseases
* Neurological diseases
* Status after actue trauma/whiplash
* Status after neoplasms in the area of the spinal column
* Acute severe comorbid mental illness or other acute severe comorbid somatic illness
* Pregnancy
* Current pension application
* Regular use of corticosteroids, opiates, muscle relaxants, or antidepressants
* Simultaneous participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-01-10 (Actual); Study Completion 2025-09-29 (Actual)

PRIMARY OUTCOMES:
Functional Impairment | Week 12
  Oswestry Disability Index (ODI): Self-report scale from 0 to 50 points with higher scores indicate higher functional impairment.

SECONDARY OUTCOMES:
Functional Impairment | Week 26
  Oswestry Disability Index (ODI): Self-report scale from 0 to 50 points with higher scores indicate higher functional impairment.
Functional Impairment | Week 52
  Oswestry Disability Index (ODI): Self-report scale from 0 to 50 points with higher scores indicate higher functional impairment.
Pain Intensity | Week 12
  Numeric rating scale (NRS): Self-report scale from 0-10 points with 0=no pain and 10=worst pain.
Pain Intensity | Week 26
  Numeric rating scale (NRS): Self-report scale from 0-10 points with 0=no pain and 10=worst pain.
Pain Intensity | Week 52
  Numeric rating scale (NRS): Self-report scale from 0-10 points with 0=no pain and 10=worst pain.
Health-related Quality of Life | Week 12
  Short Form Health Survey (SF-12): Self-report scale with two subscales (physical and mental qualityy of life). Higher scores indicate better health-related quality of life.
Health-related Quality of Life | Week 26
  Short Form Health Survey (SF-12): Self-report scale with two subscales (physical and mental qualityy of life). Higher scores indicate better health-related quality of life.
Health-related Quality of Life | Week 52
  Short Form Health Survey (SF-12): Self-report scale with two subscales (physical and mental qualityy of life). Higher scores indicate better health-related quality of life.
Severity of Depressive Symptoms | Week 12
  Center for Epidemiologic Studies Depression Scale (CES-D): 10-item self-report short form of the CES-D. Higher scores indicate higher severity of depressive symptoms.
Severity of Depressive Symptoms | Week 26
  Center for Epidemiologic Studies Depression Scale (CES-D): 10-item self-report short form of the CES-D. Higher scores indicate higher severity of depressive symptoms.
Severity of Depressive Symptoms | Week 52
  Center for Epidemiologic Studies Depression Scale (CES-D): 10-item self-report short form of the CES-D. Higher scores indicate higher severity of depressive symptoms.
Severity of Anxious Symptoms | Week 12
  Patient-Reported Outcomes Measurement Information System (PROMIS): 7-item self-report anxiety subscale. Higher scores indicate higher severity of anxious symptoms.
Severity of Anxious Symptoms | Week 26
  Patient-Reported Outcomes Measurement Information System (PROMIS): 7-item self-report anxiety subscale. Higher scores indicate higher severity of anxious symptoms.
Severity of Anxious Symptoms | Week 52
  Patient-Reported Outcomes Measurement Information System (PROMIS): 7-item self-report anxiety subscale. Higher scores indicate higher severity of anxious symptoms.
Global Improvement | Week 12
  Patient Global Impression of Improvement Scale (PGI-I): 7-point self-report scale from 1=very much improved to 7=very much worse.
Global Improvement | Week 26
  Patient Global Impression of Improvement Scale (PGI-I): 7-point self-report scale from 1=very much improved to 7=very much worse.
Global Improvement | Week 52
  Patient Global Impression of Improvement Scale (PGI-I): 7-point self-report scale from 1=very much improved to 7=very much worse.
Number of Patients with Adverse Events | Week 12
  Number of Patients with Adverse Events
Total Number (and Type) of Adverse Events | Week 12
  Total Number (and Type) of Adverse Events

OTHER OUTCOMES:
Body Awareness | Week 12
  Body Responsiveness Questionnaire (BRQ): 7-iten self-report scale with 3 subscales (Importance of Interoceptive Awareness, Perceived Connection, Suppression of Bodily Sensations). Higher scores indicate higher body awareness on the two subscales Importance of Interoceptive Awareness and Perceived Connection, while higher scores indicate lower body awareness on the subscale Suppression of Bodily Sensations.
Body Awareness | Week 26
  Body Responsiveness Questionnaire (BRQ): 7-iten self-report scale with 3 subscales (Importance of Interoceptive Awareness, Perceived Connection, Suppression of Bodily Sensations). Higher scores indicate higher body awareness on the two subscales Importance of Interoceptive Awareness and Perceived Connection, while higher scores indicate lower body awareness on the subscale Suppression of Bodily Sensations.
Body Awareness | Week 52
  Body Responsiveness Questionnaire (BRQ): 7-iten self-report scale with 3 subscales (Importance of Interoceptive Awareness, Perceived Connection, Suppression of Bodily Sensations). Higher scores indicate higher body awareness on the two subscales Importance of Interoceptive Awareness and Perceived Connection, while higher scores indicate lower body awareness on the subscale Suppression of Bodily Sensations.
Fear-related Avoidance Beliefs | Week 12
  Fear Avoidance Belief Questionnaire (FABQ): 16-item self-report scale with two subscales (fear-avoidance beliefs about physical activity and fear-avoidance beliefs about work). Higher scores indicate higher fear-avoidance beliefs.
Fear-related Avoidance Beliefs | Week 26
  Fear Avoidance Belief Questionnaire (FABQ): 16-item self-report scale with two subscales (fear-avoidance beliefs about physical activity and fear-avoidance beliefs about work). Higher scores indicate higher fear-avoidance beliefs.
Fear-related Avoidance Beliefs | Week 52
  Fear Avoidance Belief Questionnaire (FABQ): 16-item self-report scale with two subscales (fear-avoidance beliefs about physical activity and fear-avoidance beliefs about work). Higher scores indicate higher fear-avoidance beliefs.
Pain Acceptance | Week 12
  Chronic Pain Acceptance Questionnaire (CPAQ): 20-item self-report scale one sumscale and two subscales (activity engagement and pain willingness). Higher schroes indicate higher pain acceptance.
Pain Acceptance | Week 26
  Chronic Pain Acceptance Questionnaire (CPAQ): 20-item self-report scale one sumscale and two subscales (activity engagement and pain willingness). Higher schroes indicate higher pain acceptance.
Pain Acceptance | Week 52
  Chronic Pain Acceptance Questionnaire (CPAQ): 20-item self-report scale one sumscale and two subscales (activity engagement and pain willingness). Higher schroes indicate higher pain acceptance.
Use of Pain Medication | Week 1-12
  The amount of pain medication during the active study period will be assessed by Defined Daily Doses (DDD) via a diary.
Freuqnecy of Homework | Week 1-12
  The total time of performed homework (CST or PMR) during the active study period will be assessed via a diary.
Treatment Expectations | Week 1
  Treatment Credibility Scale (TCS): 1-item self-report numeric rating subscale of the TCS ("Are you confident this treatment will alleviate the pain you feel?") from 0=totally disagree to 10=totally agree. Higher scores indicate higher treamtent expectations.
Treamtent Credibility | Week 12
  Treatment Credibility Scale (TCS): 3-item self-report numeric rating subscale of the TCS from 0=totally disagree to 10=totally agree. Higher scores indicate higher treamtent credibility.
Therapist-Patient-Relationship | Week 12
  Helping Alliance Questionnaire (HAQ): 11-item self-report scale with two subscales (quality of the therapeutic relation and satisfaction with the treatment). Higher scores indicate a higher quality of the therapeutic relation / a higher satisfaction.
Interview | Week 12
  Semi-structured interview based on body image & pain drawings (at week 1 and 12)
Craniosacral-specific Quality of Life | Week 12
  Warwick Holistic Health Questionnaire (WHHQ): 25-item scale ranging from 0 to 100 points. Higher scores indicate higher craniosacral-specific quality of life.
Craniosacral-specific Quality of Life | Week 26
  Warwick Holistic Health Questionnaire (WHHQ): 25-item scale ranging from 0 to 100 points. Higher scores indicate higher craniosacral-specific quality of life.
Craniosacral-specific Quality of Life | Week 52
  Warwick Holistic Health Questionnaire (WHHQ): 25-item scale ranging from 0 to 100 points. Higher scores indicate higher craniosacral-specific quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Dobos, Prof. MD, Study Director — Center for Integrative Medicine and Planetary Health, University Hospital Essen, University of Duisburg-Essen
Locations (1):
- Center for Integrative Medicine and Planetary Health, University Hospital Essen, University of Duisburg-Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No